CLINICAL TRIAL: NCT02621671
Title: Communicating Multiple Disease Risks: A Translation of Risk Prediction Science
Brief Title: Communicating Multiple Disease Risks
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201501028
Record Dates: First submitted 2015-11-19; First posted 2015-12-03 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Healthy
Keywords: Healthy Volunteers
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Cognitive Interviews (Experimental): * Participants will complete several survey items, view 1 of 8 disease risk pictures (selected at random), and then complete further survey questions.
  * Participants will then be recorded giving their opinions on the remaining 7 disease risk pictures which depict the hypothetical risk of disease.
  * The entire visit will take no more than 90 minutes with no follow-up.
  * The first 10-20 participants will be randomized to this arm.
  Interventions: Behavioral: Cognitive interview; Other: Survey
- Arm 2: Experimental survey (Experimental): * Participants will be randomly assigned by GfK's computer to one of the 12 experimental conditions.
  * After completing questions about information seeking and physical activity, the participants will read a short scenario that describes the purpose of a risk assessment tool and ask them to imagine that they had just entered their information into such a tool.
  * Participants will see whichever risk ladder corresponds to the experimental condition to which they were assigned.
  * The hypothetical display will be consistent with a display generated for an individual whose risk profile includes risk increasing and decreasing factors, but does not engage in the recommended amount of physical activity.
  Interventions: Other: Survey

INTERVENTIONS:
Behavioral: Cognitive interview
  Arms: Arm 1: Cognitive Interviews
Other: Survey

SUMMARY:
Epidemiology seeks to improve public health by identifying risk factors for cancer and other diseases and conveying that information to relevant audiences. The audience is presumed to understand and use that information to make appropriate decisions about lifestyle behaviors and medical treatments. Yet, even though a single risk factor can affect the risk of multiple health outcomes, this information is seldom communicated to people in a way that optimizes their understanding of the importance of engaging in a single healthy behavior. Providing individuals with the ability to understand how a single behavior (obtaining sufficient physical activity) could affect their risk of developing multiple diseases could foster a more coherent and meaningful picture of the behavior's importance in reducing health risks, increase motivation and intentions to engage in the behavior, and over time improve public health.

The proposed study translates epidemiological data about five diseases that cause significant morbidity and mortality (i.e., colon cancer, breast cancer (women), heart disease, diabetes, and stroke) into a visual display that conveys individualized risk estimates in a comprehensible, meaningful, and useful way to diverse lay audiences.

ELIGIBILITY:
Inclusion Criteria:

* 30-65 years of age
* Able to read and communicate in English
* Not meeting national guidelines for aerobic physical activity (at least 150 minutes per week of moderate intensity aerobic physical activity)

Exclusion Criteria:

* Less than 30 years of age
* Older than 65 years of age
* Not able to read and communicate in English
* Meets national guidelines for aerobic physical activity (at least 150 minutes per week of moderate intensity aerobic physical activity)

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1191 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2017-06-27 (Actual); Study Completion 2017-06-27 (Actual)

PRIMARY OUTCOMES:
Test eight images/visual displays that communicate risk estimates of five diseases associated with physical activity as measured by participants understanding of the images/visual displays | Completion of accrual for Arm 1 participants (estimated to be 1 year)
  Survey questions will assess participants' cognitive and affective risk perceptions, response efficacy, perceived severity and reaction to the visual displays, health literacy and numeracy. The quantitative data will be examined using descriptive statistics (e.g., frequencies, mean, median, mode, range, interquartile range, standard deviation) to evaluate whether a potential variability problem exists (e.g., restricted range) .
Most effective combination of strategies in communicating multiple disease risk estimates (Arm 2 only) | Completion of accrual for Arm 2 participants (estimated to be 1 year)
  -Participants will be randomly assigned by computer to 1 of the 12 experimental conditions. After completing questions about information seeking and physical activity they will read a short scenario that describes the purpose of a risk assessment tool and asks them to imagine that they had just entered their information into such a tool. Participants will see whichever risk ladder corresponds to the experimental condition to which they were assigned. The hypothetical display will be consistent with a display generated for an individual whose risk profile includes risk increasing and decreasing factors, but does not engage in the recommended amount of physical activity. To increase feasibility for the display will show the risk of the diseases in the same order regardless of experimental condition. Participants will be allowed to view the display as long as they wish.

SECONDARY OUTCOMES:
Time that it takes to complete the survey that accompanies the images (Arm 1 only) | Completion of accrual for first Arm 1 participants (estimated to be 1 year)
  -Verify that there are no issues with comprehension or interpretation that can cause the survey to go longer than 20 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Erika Waters, Ph.D., M.P.H., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu